CLINICAL TRIAL: NCT06510140
Title: Interest in Combining Intraoperative ElectroEncephaloGram (EEG) With Assessment of Frailty to Predict Postoperative Delirium in Patients Aged >75 Years Undergoing Major Non-cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN482024/CHUSTE
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Post-operative Delirium
Keywords: Post-operative delirium; Frailty; General Anesthesia; Electroencephalogram; Electroencephalography; Older patients; Clinical frailty scale; Major non-cardiac surgery
MeSH Terms: conditions — Emergence Delirium; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-operative delirium (POD) arm (experimental group): Patients who present a post-operative delirium according to the 3D-CAM within 48h
  Interventions: Behavioral: Detection of the Post-operative delirium (POD)
- No Post-operative delirium (POD) arm (control group): Patients who do not present a post-operative delirium according to the 3D-CAM within 48h
  Interventions: Behavioral: Detection of the Post-operative delirium (POD)

INTERVENTIONS:
Behavioral: Detection of the Post-operative delirium (POD) — Detection of the early Post-operative delirium (POD) to assess the performance of a new composite score with pre-operative frailty, and per-operative ElectroEncephaloGram (EEG).

SUMMARY:
Post-operative delirium (POD) is known to be independently associated with pre-operative frailty, pre-operative cognitive status and per-operative ElectroEncephaloGram (EEG). However, no study has focused on the impact of these pre- and peri-operative outcomes on the prediction of Post-operative delirium (POD). Therefore, this study has been designed to assess the performance of a new score that includes pre-operative frailty, and per-operative ElectroEncephaloGram (EEG) in predicting post-operative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 75 yo or more undergoing a major non-cardiac surgery

Exclusion Criteria:

* Patients of less than 75 yo
* Cardiac surgery
* Minor surgery
* Opposition to the study protocol
* Presence of a delirium prior to the surgery

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients older than 75 yo, undergoing a major non-cardiac surgery under general anesthesia will be included.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Onset of an early Post-operative delirium (POD) | Hour : 48
  Investigation of an early Post-operative delirium (POD), with Confusion Assessment Method (CAM) criteria, 9-question test which assesses the presence, severity and fluctuation of nine clinical features of delirium, on a scale from 0 to 19. Higher scores indicate more severe delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Nory ELHADJENE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No